CLINICAL TRIAL: NCT03176043
Title: Could Thirst-triggered Self-administration of Intravenous Fluid Lead to More Rapid Rehydration Than Clinician-directed Infusion?
Brief Title: Patient Controlled Fluid Administration
Status: Unknown | Phase: Early Phase 1 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University College, London (Other)
Responsible Party: Principal Investigator, Fintan Hughes, Research Associate, University College, London
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Device Feasibility
Other Study IDs: 9339/001
Record Dates: First submitted 2017-05-30; First posted 2017-06-05 (Actual); Last update posted 2017-06-05 (Actual); Status verified 2017-06

CONDITIONS: Dehydration (Physiology); Thirst; Due to Deprivation of Water; Plasma Osmolality Increased; Hypovolemia
MeSH Terms: conditions — Dehydration; Hypovolemia

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Thirst Driven infusion (Experimental): Subjects who are self administering fluid will be instructed when (at any point in the experiment) they are experiencing thirst to request a fluid bolus with an electronic trigger. In response to this trigger the researcher will then deliver a 200ml bolus of IV fluid. After delivery of the fluid bolus, a lockout period is set for 15mins within which the researcher will not deliver another bolus in response to the trigger.
  Interventions: Procedure: IV Fluid Administration
- NICE infusion (Active Comparator): Subjects receiving standard fluid maintenance will receive a baseline infusion rate of 30 mL/kg/24hr (1.25 mL/kg/hr). In addition to this a 500 mL bolus will be delivered if any of the following clinical signs, indicating hypovolaemia, are observed on regular examination: low peripheral perfusion, heart rate >90 /min, systolic BP <100 mmHg, respiratory rate >20, peripheral capillary refill >2sec. A maximum of 2000 mL of fluid will be delivered by additional boluses.
  Interventions: Procedure: IV Fluid Administration

INTERVENTIONS:
Procedure: IV Fluid Administration — Administration of 4% Dextrose in 0.18% Sodium Chloride, through an IV cannula via a volumetric infusion pump.

SUMMARY:
The purpose of the study is to determine whether participants who are dictating their own administration of IV fluid boluses in response to thirst, receive better protection from hypovolaemia and volume overload than those who undergo routine fluid management.

Thirst is prominent in critically ill patients and is related to dehydration. In a recent study of the symptoms experience in ITU patients at high risk of dying, the sensation of thirst was reported in 70.8% of assessments made and was considered to be one of the most intense stressors. Thirst and dehydration can be combated in an ITU setting by consuming oral fluids and through administration of intravenous fluids. However, in older adults, frailty and dysphagia reduces patients' capability to access fluid and results in thirst. In addition, the administration of IV fluids is determined by the attending physician and is often only re-evaluated on a daily or twice-daily basis.

The Quench machine has been designed to allow the patient to have more control over their oral and IV fluid administration protocol. This may help reduce the sensation of thirst and dehydration in patients. The machinery is an automated fluid delivery system that will administer a given bolus of IV fluid in response to a trigger provided by the patient.

The purpose of the current study is to examine the physiological basis for the functional benefit of this Quench system by investigating the effectiveness of the thirst response in healthy humans as a guide for administration of intravenous fluid boluses.

To explore this, the investigators have designed a randomised, cross-over study. On one visit IV fluid boluses will be administered as per the participants' request in response to thirst. In the second arm of the study participants will be administered routine IV fluid maintenance as per NICE guidelines. Body mass at the end of a 4 hour fluid administration intervention will be our primary research outcome and will be compared between the two arms of the study.

From this comparison the investigators hope to show that a patient would be able to accurately manage their level of hydration, both in terms of correcting dehydration and avoiding fluid overload. It is thought that avoiding states of fluid imbalance can reduce post surgical recovery times, reduce the incidence of post operative complications and avoid critical complications of fluid imbalance, such as acute kidney injury.

DETAILED DESCRIPTION:
The purpose of the study is to investigate whether participant dictated fluid bolus administration in response to their symptom of experienced thirst is a viable basis to guide a clinical practice of fluid maintenance and correction of hydration status. To this end the experiment will compare the implementation of this fluid maintenance mechanism on volume depleted healthy participants to a program of routine fluid maintenance.

The null hypothesis is that the hydration state of the participants, as measured by change in body weight and plasma osmolality, will be no better corrected and managed by a thirst dictated management system than by routine maintenance.

The study has a cross-over design, used to ensure differences in hydration status, or lack there of, can be attributed to the methods of fluid administration in question, without differences between individuals confounding the results.

The participants will be required to attend the laboratory on two occasions for approximately 5 hours each visit, for arm A and B of the study. The two visits will be separated by 7 to 14 days. On each visit standard IV fluids will be administered The evening before each visit participants will be required to take 40mg of the water tablet called furosemide and refrain from drinking fluids. This is used in order to dehydrate the participant and reduce body mass by between 2 - 4%. The participant needs to be dehydrated in order to promote a thirst response so that the interventions can be studied in a cohort of participants representative of hypovolemic patients post surgery

On both visits an indwelling cannula will be placed into a vein in the participants' arm, to administer IV fluid on the participants' non dominant side. Before fluid administration this will be used to draw a blood sample for plasma osmolality measurements. A second blood sample with be drawn from a vein on the opposite arm following the fluid infusion.

For arm A: the participant will request the administration of 200ml boluses of IV fluid at any point that they experience thirst. This administration will be limited to one bolus every 15 minutes.

For arm B: participants will receive routine fluid maintenance as dictated by the NICE guidelines.

During both trials, low intensity exercise will be permitted (walking, standing, sitting) although high intensity exercise is not allowed. Entertainment in the form of a computer with internet access and DVDs will be provided.

The arm of the study the patient will undergo in the first week will be determined according to a randomised list. However, due to the nature of the investigation the arm of the study be undergone by the patient can not be blinded from the researchers or participant. All measurements, except the perception of thirst questioning, are objective measures, such as weight, plasma osmolality, haematocrit and blood sodium levels. This will minimise any researcher bias.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male volunteers, age range of 18-65 years weighing between 60-100 kg,

Exclusion Criteria:

* Individuals will not be allowed to take part in the study if health screening reveals any cardiovascular, respiratory, renal or metabolic disorder, or identifies any contraindication to Furosemide administration. Furthermore, individuals presenting at the laboratory with febrile symptoms will not be allowed to take part in the study until the fever subsides. During the period of study, individuals will not be allowed to take medications other than those stated in the study protocol and will be excluded if avoiding medication conflicts with previous medical advice.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Enrollment: 16 (Estimated)
Dates: Start 2016-08-01 (Actual); Primary Completion 2017-08 (Estimated); Study Completion 2017-08 (Estimated)

PRIMARY OUTCOMES:
Volume of Fluid Administered | 4 hours
  Volume of Fluid Administered, this total volume measured in ml will be logged by the volumetric pump.

SECONDARY OUTCOMES:
Change in body mass | 4 hours
  Change in body mass from the beginning to the end of each infusion. Measured as the subject stands on an electronic scale. Any urine output will we weighed in containers and added to the final mass.
Change in urine specific gravity | 4 hours
  Change in urine specific gravity from the beginning to the end of each infusion. Urine samples taken at the beginning of the study and at the end (subjects having emptied their bladders 30 minutes prior) will be dipped to measure specific gravity.
Change in plasma osmolality | 4 hours
  Change in plasma osmolality in the blood samples drawn at the beginning and end of each infusion. Samples will be centrifuged before being analysed by freezing point depression.

CONTACTS AND LOCATIONS:
Locations (1):
- Institute of Sport Exercise & Health, London, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hughes F, Ng SC, Mythen M, Montgomery H. Could patient-controlled thirst-driven fluid administration lead to more rapid rehydration than clinician-directed fluid management? An early feasibility study. Br J Anaesth. 2018 Feb;120(2):284-290. doi: 10.1016/j.bja.2017.11.077. Epub 2017 Dec 2. PMID 29406177